CLINICAL TRIAL: NCT07051642
Title: The Dino Study: Rationale and Study Protocol for a Randomized Controlled Trial Evaluating the Incredible Years Dinosaur Program With Daily Assessments
Brief Title: Dino Study: Daily Intervention-based Research on Nurturing Opportunities in Young Children
Acronym: Dino
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Rabia Chhangur, Dr., Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSB_RP2172; 406.XS.24.03.088 (Other Grant/Funding Number: Netherlands Organisation for Scientific Research)
Record Dates: First submitted 2025-06-25; First posted 2025-07-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Behavior Problems in Children; Parent-Child Relations; Oppositional Behavior; Social Skills
Keywords: Incredible Years Dinosaur Program; Conduct problems; Emotional sensitivity; Parent-child interaction; Daily diary; Experience Sampling Method; Randomized controlled trial; Behavioral intervention
MeSH Terms: conditions — Social Skills; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Participants (children aged 4-8 years and one parent per family) are randomly assigned (1:1) to either the intervention group, which receives the Incredible Years Dinosaur Program, or a waitlist control group. Both groups are assessed at baseline and after the 18-week study period. The waitlist group receives the intervention after the final assessment but is not included in the intervention analysis.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded trial in which the outcomes assessors (e.g., coders) are unaware of participant group allocation. Participants, parents, and group leaders are not blinded due to the nature of the behavioral intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incredible Years Dinosaur Program (Experimental): Children in this arm will participate in the Incredible Years Small Group Dinosaur Child Program, a structured, evidence-based behavioral intervention designed for children aged 4-8 with conduct problems. The program consists of 18 weekly sessions of approximately two hours each, delivered in small groups by certified trainers. The sessions use play-based activities (e.g., puppets, storytelling, role-play) to promote emotional regulation, prosocial behavior, and problem-solving skills.
  Interventions: Behavioral: Incredible Years Dinosaur Child Program
- Waitlist Control Group (No Intervention): Children in this arm will not receive any structured intervention during the 18-week study period but will continue to access usual care or services as needed. After completing the post-intervention assessment, they will be offered the Incredible Years Dinosaur Program outside of the research context, on a voluntary basis.

INTERVENTIONS:
Behavioral: Incredible Years Dinosaur Child Program — The Incredible Years Dinosaur Child Program is a structured, manualized group intervention designed for children aged 4 to 8 years with elevated or (sub)clinical conduct problems. The program consists of 18 weekly group sessions lasting approximately two hours each. Sessions are delivered in small groups (5-6 children per group) by certified trainers and follow a developmentally appropriate, play-based curriculum. Intervention components include storytelling with puppets, role-play, video modeling, and group discussions. The program aims to enhance emotional regulation, social competence, and problem-solving skills. The Dutch version of the program is used in this study and implemented in both clinical and preventive settings.
  Arms: Incredible Years Dinosaur Program

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the Incredible Years Dinosaur Program in children aged 4 to 8 years with conduct problems. The main questions it aims to answer are:

* Does participation in the Dinosaur Child Program lead to greater improvements in children's emotional, social, and cognitive functioning, and reductions in externalizing behavior compared to a waitlist control group?
* Does the intervention reduce emotional variability and daily behavior problems as captured through daily diary assessments?
* Does the intervention improve daily parent-child dynamics, including reduced emotional escalation and more shared positive affect?

Researchers will compare children in the intervention group to those in the waitlist control group to see if the program leads to better emotional regulation, fewer behavior problems, and improved parent-child interactions.

Participants will:

* Be randomly assigned to either the intervention or waitlist control group (1:1) Receive 18 weekly small-group sessions (if in the intervention condition) using the Incredible Years Dinosaur Program
* Complete daily diaries with their parent using the m-Path app during a 20-week period (baseline, intervention, follow-up)
* Complete standardized pre- and post-intervention assessments via parent, teacher, and child reports

DETAILED DESCRIPTION:
The Dino Study is a two-arm randomized controlled trial (RCT) designed to evaluate the effectiveness of the Incredible Years (IY) Small Group Dinosaur Child Program in young children (ages 4 to 8) with elevated or (sub)clinical levels of conduct problems. Conduct problems at this age are associated with long-term risks for poor academic, social, and mental health outcomes, yet current interventions rarely account for individual differences in children's emotional responsiveness and daily functioning. This study introduces the Dinosaur Program in the Netherlands and combines conventional pre- and post-intervention assessments with an intensive longitudinal diary design to examine both group-level effects and intra-individual mechanisms of change.

A total of 120 children and one parent per family will be recruited through partnerships with primary schools and mental health organizations. Families are eligible if the child is aged 4 to 8 years, has sufficient Dutch language skills, and shares daily contact with the participating caregiver. Children with an intellectual disability (IQ < 70) or insufficient Dutch fluency will be excluded. After informed consent, families will be randomly allocated (1:1) to either the intervention or waitlist control condition. The intervention group will participate in 18 weekly 2-hour group sessions delivered by certified IY group leaders. The waitlist group receives care-as-usual and is offered the intervention after the posttest.

The Incredible Years Dinosaur Child Program is a structured, manualized group intervention based on cognitive-behavioral principles. It aims to enhance emotional regulation, prosocial behavior, and problem-solving abilities through playful, developmentally appropriate activities such as puppet play, role-play, group discussion, and storytelling. While parents do not receive formal training, they are indirectly exposed to program content through letters and reading assignments. The program has been widely implemented and evaluated internationally, but this study is the first to integrate it with daily diary methods to capture day-to-day variability in children's behavior and parent-child dynamics.

Primary outcomes focus on externalizing behavior, cognitive and social-emotional functioning, assessed via standardized parent, teacher, and child instruments. Secondary outcomes are derived from daily diaries and capture fluctuations in emotions, behavior, and dyadic emotional exchanges. Daily assessments will be collected using the m-Path app, completed jointly by parent and child every evening over a 20-week period (1 week baseline, 18 weeks intervention, 1 week follow-up). This approach enables fine-grained modeling of emotional variability and relational processes in the child's natural environment.

The study is informed by the Environmental Sensitivity Framework, which posits that children vary in their responsiveness to environmental input. Emotional sensitivity will be operationalized as moment-to-moment fluctuations in daily negative affect prior to the intervention. Multilevel and time-series analyses will be used to evaluate overall treatment effects as well as dynamic, intra-individual change patterns. Key hypotheses include: (1) children in the intervention group will show greater improvements in externalizing behavior and social functioning than those in the control group; (2) daily negative affect and behavior problems will decline more in the intervention group; and (3) intervention effects will be moderated by children's baseline emotional sensitivity.

Findings will contribute to the emerging field of precision prevention by identifying which children benefit most from structured group interventions and under what conditions. The integration of Intensive Longitudinal Data (ILD )with a randomized trial design allows for a mechanistic, personalized understanding of behavioral change in young children and their families.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 8 years
* At least one parent or primary caregiver willing and able to participate in the study and complete daily diary assessments
* Sufficient Dutch language proficiency in child and parent to complete questionnaires and daily diary reports
* Parental indication that the child shows elevated or (sub)clinical levels of conduct problems in daily life (e.g., frequent defiance, aggression, or rule- breaking behavior

Exclusion Criteria:

* Intellectual disability in the child (IQ < 70)
* Child lives primarily in a different household during weekdays (e.g., institutional care, full-time co-parenting arrangement)
* Parent/child does not have sufficient Dutch language proficiency

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in social competence (parent-reported and teacher-reported) | Baseline (T1) to Post-Intervention (T2); ~19 weeks
  The Parent version (P-COMP) completed by parents The Teacher version (T-COMP) completed by teachers Both versions include items assessing prosocial behavior, cooperation, empathy, and emotional self-regulation. Scores from baseline (T1) and post-intervention (T2) will be compared to evaluate changes in social functioning across home and school contexts.
Change in externalizing behavior (parent-reported and teacher-reported) | Baseline (T1) to Post-Intervention (T2); ~19 weeks
  Externalizing behavior will be assessed using standardized instruments at two time points:
  The Eyeberg Child Behavior Inventory (ECBI) and Child Behavior Checklist (CBCL) completed by parents, and The Teacher's Report Form (c-TRF/TRF) completed by teachers. Both instruments are part of the Achenbach System of Empirically Based Assessment (ASEBA) and include subscales measuring aggressive and rule-breaking behavior. The primary outcome is the change in externalizing scores from baseline (T1) to post-intervention (T2), approximately 19 weeks apart.
Change in executive functioning (parent-reported and teacher-reported) | Baseline (T1) to Post-Intervention (T2); ~19 weeks
  Executive functioning will be measured with the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2). The Parent Form (60 items) and Teacher Form (61 items) use a 3-point Likert scale (1 = never, 2 = sometimes, 3 = often) to rate everyday behaviors reflecting executive skills (for example, "Has trouble remembering things, even for a few minutes"). For this study the Global Executive Composite (GEC) will serve as the primary outcome. GEC scores from baseline (T1) and post-intervention (T2) will be compared to evaluate changes in children's executive functioning across home and school contexts.
Change in child language and communication behavior (parent-reported) | Baseline (T1) to Post-Intervention (T2); ~19 weeks
  Child language and communication functioning will be assessed using the Children's Communication Checklist - Second Edition, Dutch version (CCC-2-NL). This 70-item parent-report questionnaire covers both structural language skills (e.g., syntax, semantics) and pragmatic communication abilities (e.g., inappropriate initiation, use of context, nonverbal communication). Each item is rated on a 4-point scale (0 = "less than once a week or never" to 3 = "several times a day or always"). The General Communication Composite (GCC) will be used as the primary outcome measure to evaluate change in communicative functioning from baseline (T1) to post-intervention (T2).
Change in child-assessed emotional understanding and problem-solving skills | Baseline (T1) to Post-Intervention (T2); ~19 weeks
  Children's emotional understanding and problem-solving skills will be assessed using two structured, age-appropriate tasks:
  The Wally Feeling Test, which measures the child's ability to recognize and explain emotional expressions in cartoon-based vignettes.
  The Wally Problem Solving Test, which presents illustrated social dilemmas and asks children to generate possible solutions.
  Responses are coded for emotional awareness, perspective-taking, and cognitive flexibility. Change from baseline (T1) to post-intervention (T2) will be evaluated to determine the impact of the intervention on child-level socio-emotional competencies.

SECONDARY OUTCOMES:
Daily dynamic emotional processes (ESM-based) | Daily over 20 weeks
  This outcome captures children's daily emotional instability and problem-solving behaviors, measured using parent-child dyadic reports via the m-Path mobile app. Emotional instability is defined as within-person fluctuations in negative affect (e.g., anger, sadness), while coping is operationalized as the use of emotion regulation strategies reported by the child. These indicators are collected daily to examine how children's emotional self-regulation develops over the course of the intervention.
Daily behavioral processes within families (Dyadic ESM-based) | Daily over 20 weeks
  This outcome captures parent-child affective dynamics in daily life, based on separate reports from parents and children. Negative interactions are assessed through measures of emotional escalation, conflict, and anger. Positive interactions include shared emotional moments and expressions of warmth. These data allow for analysis of affective synchrony, divergence, and co-regulation over time, reflecting how the intervention impacts relationship quality.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy considerations involving young children and their families. The data include sensitive mental health and behavioral information, and participants did not consent to public data sharing.

REFERENCES:
- [Background] Webster-Stratton C, Reid J, Hammond M. Social skills and problem-solving training for children with early-onset conduct problems: who benefits? J Child Psychol Psychiatry. 2001 Oct;42(7):943-52. doi: 10.1111/1469-7610.00790. PMID 11693589
- [Background] Webster-Stratton C, Jamila Reid M, Stoolmiller M. Preventing conduct problems and improving school readiness: evaluation of the Incredible Years Teacher and Child Training Programs in high-risk schools. J Child Psychol Psychiatry. 2008 May;49(5):471-88. doi: 10.1111/j.1469-7610.2007.01861.x. Epub 2008 Jan 21. PMID 18221346
- [Derived] Chhangur RR, Smalle EHM, Dejonckheere E, van der Zwaag G. The Dino Study: Rationale and protocol for a randomized controlled trial of the Incredible Years Dinosaur Program with daily assessments. PLoS One. 2025 Sep 8;20(9):e0330597. doi: 10.1371/journal.pone.0330597. eCollection 2025. PMID 40920805